CLINICAL TRIAL: NCT03805126
Title: Expanding the UTHealth Medical Legal Partnership to Improve Mental Health for Low-Income Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Medical Center Foundation (Unknown); University of Houston (Other); William Marsh Rice University (Other)
Responsible Party: Principal Investigator, Winston Liaw, Associate professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-18-1037
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Health-harming Legal Needs

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Legal Partnership (Experimental): With the medical legal partnership, lawyers are embedded in clinics, and lawyers consult with patients who are identified as having health-harming legal needs (HHLNs). This arm will also receive usual care, which includes consultation with a social worker and a community health worker.
  Interventions: Behavioral: Medical Legal Partnership; Behavioral: Usual Care
- Usual Care (Active Comparator): Usual care includes consultation with a social worker and a community health worker.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Medical Legal Partnership — With the medical legal partnership, lawyers are embedded in clinics, and lawyers consult with patients who are identified as having health-harming legal needs (HHLNs). This arm will also receive usual care, which includes consultation with a social worker and a community health worker.
  Arms: Medical Legal Partnership
Behavioral: Usual Care — Usual care includes consultation with a social worker and a community health worker.

SUMMARY:
The aim of this study is to test whether participation of low-income patients with health-harming legal needs (HHLNs) in a medical legal partnership (MLP) results in improved mental health, improved quality of life, reduced utilization, and increased resolution of HHLNs.

ELIGIBILITY:
Inclusion Criteria:

* low-income individuals (Low-income is defined as earning less than 200% of the Federal Poverty Level)
* individuals with HHLNs
* English or Spanish speaking

Exclusion Criteria:

* self-identified as being at significant and immediate risk due to HHLNs (e.g., a situation that involves imminent risk to the patient such as domestic violence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Stress as assessed by the Perceived Stress Scale | baseline
  The perceived stress scale consists of 10 items, with each item ranging from 0-4, for a total score range of 0-40. A higher score indicates a worse outcome.
Stress as assessed by the Perceived Stress Scale | 3 months
  The perceived stress scale consists of 10 items, with each item ranging from 0-4, for a total score range of 0-40. A higher score indicates a worse outcome.
Stress as assessed by the Perceived Stress Scale | 6 months
  The perceived stress scale consists of 10 items, with each item ranging from 0-4, for a total score range of 0-40. A higher score indicates a worse outcome.
Stress as assessed by the Perceived Stress Scale | 12 months
  The perceived stress scale consists of 10 items, with each item ranging from 0-4, for a total score range of 0-40. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Anxiety as assessed by the Generalized Anxiety Disorder 7-item scale | baseline
  The Generalized Anxiety Disorder scale consists of 7 items, with each item ranging from 0-3, for a total score range of 0-21. A higher score indicates a worse outcome.
Anxiety as assessed by the Generalized Anxiety Disorder 7-item scale | 3 months
  The Generalized Anxiety Disorder scale consists of 7 items, with each item ranging from 0-3, for a total score range of 0-21. A higher score indicates a worse outcome.
Anxiety as assessed by the Generalized Anxiety Disorder 7-item scale | 6 months
  The Generalized Anxiety Disorder scale consists of 7 items, with each item ranging from 0-3, for a total score range of 0-21. A higher score indicates a worse outcome.
Anxiety as assessed by the Generalized Anxiety Disorder 7-item scale | 12 months
  The Generalized Anxiety Disorder scale consists of 7 items, with each item ranging from 0-3, for a total score range of 0-21. A higher score indicates a worse outcome.
Depression as assessed by the Center for Epidemiologic Studies Depression Scale | baseline
  The Center for Epidemiologic Studies Depression Scale consists of 20 items, with each item ranging from 0-3, for a total score range of 0-60. A higher score indicates a worse outcome.
Depression as assessed by the Center for Epidemiologic Studies Depression Scale | 3 months
  The Center for Epidemiologic Studies Depression Scale consists of 20 items, with each item ranging from 0-3, for a total score range of 0-60. A higher score indicates a worse outcome.
Depression as assessed by the Center for Epidemiologic Studies Depression Scale | 6 months
  The Center for Epidemiologic Studies Depression Scale consists of 20 items, with each item ranging from 0-3, for a total score range of 0-60. A higher score indicates a worse outcome.
Depression as assessed by the Center for Epidemiologic Studies Depression Scale | 12 months
  The Center for Epidemiologic Studies Depression Scale consists of 20 items, with each item ranging from 0-3, for a total score range of 0-60. A higher score indicates a worse outcome.
Quality of life as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) | baseline
  The Patient-Reported Outcomes Measurement Information System (PROMIS) consists of 29 items, with 28 of the items ranging from 1-5 and 1 item ranging from 0-10, for a total score range of 28-150. A higher score indicates a worse outcome.
Quality of life as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) | 3 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) consists of 29 items, with 28 of the items ranging from 1-5 and 1 item ranging from 0-10, for a total score range of 28-150. A higher score indicates a worse outcome.
Quality of life as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) | 6 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) consists of 29 items, with 28 of the items ranging from 1-5 and 1 item ranging from 0-10, for a total score range of 28-150. A higher score indicates a worse outcome.
Quality of life as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) | 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) consists of 29 items, with 28 of the items ranging from 1-5 and 1 item ranging from 0-10, for a total score range of 28-150. A higher score indicates a worse outcome.
Number of Urgent Care Visits | baseline
Number of Urgent Care Visits | 3 months
Number of Urgent Care Visits | 6 months
Number of Urgent Care Visits | 12 months
Number of Emergency Department Visits | baseline
Number of Emergency Department Visits | 3 months
Number of Emergency Department Visits | 6 months
Number of Emergency Department Visits | 12 months
Number of Hospital Visits | baseline
Number of Hospital Visits | 3 months
Number of Hospital Visits | 6 months
Number of Hospital Visits | 12 months
Percentage of baseline health-harming legal needs that were resolved | baseline
Percentage of baseline health-harming legal needs that were resolved | 3 months
Percentage of baseline health-harming legal needs that were resolved | 6 months
Percentage of baseline health-harming legal needs that were resolved | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Winston Liaw, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Jensen Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liaw W, Northrup TF, Stotts AL, Bakos-Block C, Suchting R, Chen A, Hernandez A, Finzetto L, Green C, Murphy T. Medical-Legal Partnership Effects on Mental Health, Health Care Use, and Quality of Life in Primary Care: A Randomized Clinical Trial. J Am Board Fam Med. 2023 May 8;36(3):414-424. doi: 10.3122/jabfm.2022.220349R1. Epub 2023 Apr 7. PMID 37028914